CLINICAL TRIAL: NCT03120117
Title: Importance of Patient Positioning at Cough Test When Considering Success Following Sling Procedures
Acronym: DISST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michigan Institution of Women's Health PC (Other)
Responsible Party: Principal Investigator, Salil Khandwala MD, Medical Director, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIWH13-001
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Midurethral Slings
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cough Test following Sling Surgery (Experimental): All subjects enrolled will undergo sling surgery for treatment of stress urinary incontinence and subsequently asked to do a standing cough test.
  Interventions: Procedure: Cough Test following Sling Surgery

INTERVENTIONS:
Procedure: Cough Test following Sling Surgery — Enrolled subjects will undergo sling surgery who present with stress-dominated urinary incontinence. While in the operating room, the subject will be asked to stand and cough to determine if there is still leakage once the sling has been placed.
  Other Names: DISST Procedure

SUMMARY:
This is a prospective study to assess the feasibility and success of performing an intra-operative standing cough test and the correlation with the long term success of the sling surgery.

DETAILED DESCRIPTION:
The goal is to seek correlation or disparity between the supine versus the sitting cough test, supine (lying down) versus standing cough test and sitting versus the standing cough test performed at a constant bladder volume; empty in the office and full in the operating room. Secondary objective is to test if the intra-operative standing cough test at fullness correlates with long term success of the sling surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with stress-dominant urinary incontinence
* Patients who have undergone a stress test documentation both in the supine and standing/sitting position.
* Patients who have completed child bearing.
* Patients between 21 and 89 years of age.

Exclusion Criteria:

* Patients who do not agree to participate and do not sign the informed consent.
* Patients undergoing concomitant surgery
* Patients undergoing surgery under anesthesia.

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who present with recurrence of stress incontinence following sling surgery as assessed by post-operative cough test. | Within first two years following sling procedure
  Success criteria will be defined through the examination of patient's post-operative visits regarding cough stress tests in supine, sitting and standing positions where the bladder is at 10% of urodynamic fullness. Failure to meet this criteria will be considered recurrence of stress incontinence.
Number of patients who present with recurrence of stress incontinence following sling surgery as assessed by post-operative MESA questionnaire. | Within first two years following sling procedure
  Success criteria is also defined through the examination of patient's response to Medical Epidemiologic and Social Aspects of Aging 12 (MESA) to determine recurrence of stress incontinence. Failure to meet this criteria will be considered recurrence of stress incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Salil Khandwala, MD, Principal Investigator — Michigan Institute of Women's Health
Locations (1):
- Advanced Urogynecology of Michigan, P.C., Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No